CLINICAL TRIAL: NCT03809793
Title: Can the Health Benefits of a Walking-based Exercise Programme be Enhanced by Co-ingestion of a Lipid-lowering Drug?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Diabetes UK (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); Royal Liverpool University Hospital (Other Government)
Responsible Party: Principal Investigator, Jennifer Barrett, PhD researcher in Exercise Metabolism, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 250408
Record Dates: First submitted 2019-01-07; First posted 2019-01-18 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Resistance Training; acipimox

STUDY DESIGN:
Intervention Model Description: 34 pre-diabetics will be split into 2 groups; one will ingest Acipimox for 12-weeks and the other will ingest nothing.
Masking Description: both participants and investigators will know if they are ingesting Acipimox or nothing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acipimox ingestion (Active Comparator): Individuals in this group will undergo pre-assessments for body composition (DXA), Insulin sensitivity (Hyperinsulinaemic Euglycaemic clamp and continuous glucose monitor), muscle biopsies pre- and post- clamp for analysis of lipid metabolites, liver fat (MRI) and exercise capacity (VO2 max). Participants will then ingest 250 mg of Acipimox 1 hour before each exercise session of the 12 week intervention.
  Interventions: Other: Exercise Program; Diagnostic Test: DXA; Diagnostic Test: MRI; Diagnostic Test: Hyperinsulinaemic Euglycaemic Clamp; Diagnostic Test: VO2 Max; Diagnostic Test: Continuous Glucose Monitor; Procedure: Muscle Biopsies; Drug: Acipimox 250 MG
- No drug (Placebo Comparator): Individuals in this group will undergo pre-assessments for body composition (DXA), Insulin sensitivity (Hyperinsulinaemic Euglycaemic clamp and continuous glucose monitor) with muscle biopsies pre- and post- clamp for analysis of lipid metabolites, liver fat (MRI) and exercise capacity (VO2 max). Participants will then ingest nothing prior to their exercise sessions during the 12-week exercise programme.
  Interventions: Other: Exercise Program; Diagnostic Test: DXA; Diagnostic Test: MRI; Diagnostic Test: Hyperinsulinaemic Euglycaemic Clamp; Diagnostic Test: VO2 Max; Diagnostic Test: Continuous Glucose Monitor; Procedure: Muscle Biopsies

INTERVENTIONS:
Other: Exercise Program — 12-week walking based intervention (3 sessions per week)
Diagnostic Test: DXA — Participants will undergo an assessment of body composition (DXA)
Diagnostic Test: MRI — used to measure fat stored in the liver
Diagnostic Test: Hyperinsulinaemic Euglycaemic Clamp — Participants will arrive at the laboratory after an overnight fast (>10 h) to undergo a Hyperinsulinaemic euglycaemic clamp to assess whole-body insulin sensitivity. Plasma glucose will be measured at regular intervals and muscle biopsies will be obtained from the vastus lateralis muscle of one leg before and after 2 hours of the clamp.
Diagnostic Test: VO2 Max — Assessment of maximum aerobic capacity.
Diagnostic Test: Continuous Glucose Monitor — CGM sensor will be inserted to measure insulin sensitivity over a 24hr period.
Procedure: Muscle Biopsies — Participants will undergo muscle biopsies pre and post the hyperinsulinemic euglyceamic clamp from the vastus lateralis.
Drug: Acipimox 250 MG — Participants will be randomised into two groups. One group will be prescribed Acipimox that will be taken 1 hour prior to each exercise session. The other group will take no drug.
  Arms: Acipimox ingestion

SUMMARY:
Study investigates the hypothesis that an exercise programme of steady walking will have larger effects on insulin sensitivity and glycemic control when combined with Acipimox intake prior to each exercise session in people with pre-diabetes. Thirty-four sedentary, overweight/obese people (aged 25-50 years, BMI >28 kg.m-2) with pre-diabetes will be recruited using the same strategy as study 2 and split into two groups (detailed below). Participants will undergo several pre- intervention assessments, followed by a 12-week walking based intervention combined with either Acipimox ingestion or no drug ingestion, pre- each exercise session. Following this, the post-assessment measures will identical to the pre-assessment measures.

DETAILED DESCRIPTION:
Study 3 investigates the hypothesis that an exercise programme of steady walking will have larger effects on insulin sensitivity and glycaemic control when combined with Acipimox intake prior to each exercise session in people with prediabetes. Thirty-four sedentary, overweight/obese people (aged 25-50 years, BMI >28 kg.m-2) with prediabetes will be recruited using the same strategy as study 2 and split into two groups (detailed below).

Pre-intervention assessments:

Visit 1: Participants will undergo an assessment of body composition (DXA) and undertake a graded treadmill walking test to estimate maximal aerobic fitness (VO2max).

Visit 2: Participants will be able to opt to undergo an MRI scan, taking place before breakfast. The MRI scan is used to measure fat stored in the liver and muscles. A continuous glucose monitoring (CGM) sensor will be inserted to measure insulin sensitivity.

Visit 3: Participants will arrive at the laboratory after an overnight fast (>10 h) to undergo a Hyperinsulinaemic euglycaemic clamp to assess whole-body insulin sensitivity. Plasma glucose will be measured at regular intervals and muscle biopsies will be obtained from the vastus lateralis muscle of one leg before and after 2 hours of the clamp.

Exercise intervention: Pairs of participants from each group (matched for gender, age and VO2max) will be randomized to undertake 12 weeks of steady walking combined with ingestion of either Acipimox or placebo in a counter-balanced, double-blind design. Supervised treadmill walking sessions will be undertaken at LJMU three times per week, with exercise performed at a speed equivalent to 45% VO2max. Participants will initially exercise for 30 mins per session (weeks 1 and 2), and each session will increase in duration by 5 mins every 2 weeks thereafter, up to 50 minutes of exercise. 1 hour before each walking session, participants will ingest either 250 mg Acipimox or nothing.

Post-intervention assessments: The post-intervention assessments will be identical in all respects to the pre-intervention assessments and will be commenced ≥72 hours after the final training session.

ELIGIBILITY:
Inclusion Criteria:

* BMI >28 kg.m-2
* Pre-diabetic
* Not currently using any anti-diabetes medication
* Physically inactive (performing less than two 30 min structured exercise sessions per week for the last year)
* Not pregnant or currently breast feeding
* Pre-menopausal
* Not currently involved in a weight loss programme or using weight loss medication

Exclusion Criteria:

* Involved in regular exercise (engaged in more than 2 sessions of structured exercise of >30 min per week)
* Currently using anti-diabetes medication (e.g. insulin, metformin)
* Currently using niacin/vitamin B3 supplements
* Pregnant or breast feeding
* Currently engaged in active weight loss programme or using weight loss medication
* Diagnosed with chronic kidney disease

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | A change in insulin sensitivity from baseline will be compared to week 12.
  A pre- and post- hyperinsulinaemic euglycaemic clamp will assess changes in whole body insulin sensitivity.

SECONDARY OUTCOMES:
Sub-maximal VO2 walking test | A change in aerobic capacity (VO2) from baseline will be compared to week 12.
  Participants will be assessed for pre- and post- maximal aerobic capacity.
Percentage of Liver Fat | The change percentage of liver fat will be measured at baseline and be compared to value at the end of week 12.
  A pre- and post- intervention MRI scan will show any changes in Liver Fat
Changes in Intramuscular GLUT4 | A change in the co-localisation of GLUT4 will be assessed from the values from the clamp at baseline, to the clamp at week 12 after the intervention.
  Muscle biopsy samples will undergo analysis of mechanisms for insulin sensitivity and lipid metabolites using confocal immunofluorescence microscopy.
Change in intramuscular DAGs | A change in the amount of DAGs will be assessed from the values from the clamp at baseline, to the clamp at week 12 after the intervention.
  The amount of DAGs within the muscle will be analysed using liquid chromatography-mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer s Barrett, PhD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No